CLINICAL TRIAL: NCT01554449
Title: Effect of Early Upper Arm Rehabilitation After Stroke Using Adaptative Video Games
Brief Title: Upper Arm Reahabilitation After Stroke and Video Game
Acronym: MARGAUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8642; 2010-A00596-33 (Other: ID RCB)
Record Dates: First submitted 2012-03-07; First posted 2012-03-15 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Stroke; Cerebro-vascular Accident; Upper Arm Disability; Reaching; Grasping
Keywords: Stroke; Upper arm; Rehabilitation; Motor function; Video games; Virtual reality; Occupational Therapy; Functional MRI
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Serious game (Experimental): In this group, patients will have a session of conventional retraining with a serious game retraining.
  Interventions: Procedure: serious game reeducation; Procedure: functional MRI
- control patients (Active Comparator): In this group, patients will have the conventional retraining with an other conventional retrainning session. The difference between both groups of patients is the serious game session for one group and conventional session for the other group
  Interventions: Procedure: serious game reeducation; Procedure: functional MRI
- controls (Placebo Comparator): For the neurologic assessments, patients are compared to healthy patient (without stroke)
  Interventions: Procedure: functional MRI

INTERVENTIONS:
Procedure: serious game reeducation — It's a daily session (45 minutes) of reeducation by serious game (kinect) compared to a daily session (45 minutes) of conventional reeducation
  Arms: Serious game; control patients
Procedure: functional MRI — the functional MRI (siemens) will be done on 25 stroke patients and 12 healthy volunteers at baseline and at 6 weeks.

SUMMARY:
The purpose of this study is to assess the efficiency of occupational therapy enhanced by "dedicated adaptative video games" in rehabilitation of the upper arm of stroke patients in the acute phase after their cerebro-vascular accident. Our hypothesis is that occupational therapy enhanced by dedicated adaptative video games is more efficient in improving motor recovery of the upper arm than conventional occupational therapy alone.

DETAILED DESCRIPTION:
Introduction : Stroke constitutes one of the most disabiliting desease in industrialized countries, leading to major deficiencies, especially in the upper arm (concerning 50 to 80% of post-stroke patients). Upper arm rehabilitation after stroke improved during the last ten years, with the development of new rehabilitation methods including constraint induced therapy, mirror therapy, mental imaging, virtual reality and robotics. Video games and virtual reality are very promising in this field, and the development of new adaptative games dedicated to upper arm rehabilitation after stroke is necessary to enhance the benefit of those devices in therms of sensori-motor and functional recovery.

Objectives: To prove the efficiency of video-gaming (using dedicated adaptative games) on recovery of motor function of the upper armafter stroke, compared to a "conventional" rehabilitation program.

Design: Multicentric Randomized Controlled TrialParticipants: 50 early stroke patients and 12 healthy control persons will be included in this trial. Inclusion criteria for patients are as follow: age>18, onset of stroke <6 weeks, first unique supra-tentorial ischemic or haemorrhagic stroke, Fugl Meyer score of the upper arm < 30/66 at inclusion. Exclusion criteria are as follow: severe neglect or aphasia, upper arm severe orthopedic limitation, shoulder pain > 5/10, contra-indication to MRI.

Methods:All patient will get a "standard program" of rehabilitation 5 days/week duiong six weeks, including physiotherapy (one or two sessions/day), occupational therapy (one session/day) and speech therapy if necessary (one session/day). Patients will be randomized in two groups: the "treated group" receiving an additional session of 30 to 45 minutes of daily rehabilitation with video games under the supervision of an occupational therapist, and the "control group" receiving the same anount of "standard rehabilitation" provided by an occupational therapist.Assesment will be conducted at inclusion (J0), at the end of the program (Week 6: W6) and at follow-up (end of month 6: M6)).

Recorded datas: The primary endpoint is the difference in increasing the upper arm Fugl Meyer Score (FMS) between both groups at W6. Secondary criterions include: FMS at M6, Box and Block Test at W6 and M6, Nine Hole Peg test at W6 and M6, Wolf Motor Function Test at W6 and M6, Motor Activity Log at W6 and M6, Barthel Index at W6 and M6, SF-36 at W6 and M6. Functional MRI and tensor diffusion imaging will also be conducted in 25 patients and 12 controls, at J0 and W6. Evolution of cerebral plasticity and correlations between cerebral re-organisations and kinematic characteristics of upper arm movements will be provided.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* onset of stroke < 6 weeks
* first unique supra-tentorial ischemic or haemorhagic stroke
* Fugl Meyer score of the upper arm < 30/66 at baseline

Exclusion Criteria:

* severe neglect or aphasia
* upper arm severe orthopedic limitation
* shoulder pain > 5/10
* pregnancy < 3 months
* Contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-09-12 (Actual); Primary Completion 2016-03-22 (Actual); Study Completion 2016-07-12 (Actual)

PRIMARY OUTCOMES:
Efficacy assessment of the serious game on the recovery of the upper limb | at 6 weeks
  Difference in increase of the Upper Arm Fugl Meyer Score (max: 66) between both groups, at the end of the rehabilitation program (week 6)

SECONDARY OUTCOMES:
Fugl Meyer Score between both groups | at 6 Months
  Difference in increase of the Upper Arm Fugl Meyer Score (max: 66) between both groups, at the end of the study(6 months)
Box and Block Test assessment between both groups | at 6 Weeks and 6 Months
  The box and block test assess the global capacities of prehension of patients. It's important to compare these capacities between both groups of treatment.
Wolf Motor Function Test assessment between both groups. | at 6 weeks and at 6 months
  To assess the motor capacity by the Wolf motor funtion at 6 Weeks and after 6 Months.
Motor Activity Log assessment between both groups | at 6 weeks and at 6 months
  This test assess the frequency of use and the quality of the movement.
Barthel Index and SF-36 | at 6 weeks and at 6 months
  The Barthel Index assess the global functional capacities by a score (calculated /100)between both groups of patients. The SF-36 is a self-questionnaire which permits the evalulation of quality of life.
Functional MRI Assessment between controls and patients | at baseline and at 6 weeks
  Functional MRI permits to study of the topographics neuronal circuits involved in the recovery of the motor functions of the upper limb: evaluation of the profiles of activation involved in the execution of the movement of fingers flexion / extension involving the right hemisphere and then the left hemisphere.
Nine Hole Peg test assessment between both groups | at 6 weeks and at 6 months
  To assess the efficacy of Serious Game on manual dexterity on the duration of Nine Hole Peg test.
tensor diffusion analysis between controls and patients | at 6 weeks
  The tensor diffusion imaging will also be conducted in 25 patients and 12 controls, at baseline and at 6 weeks. Evolution of cerebral plasticity and correlations between cerebral re-organisations and kinematic characteristics of upper arm movements will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Laffont Isabelle, MD, PhD, Principal Investigator — CHRU de Montpellier
Locations (1):
- CHRU de Montpellier, Montpellier, France

REFERENCES:
- [Derived] Laffont I, Froger J, Jourdan C, Bakhti K, van Dokkum LEH, Gouaich A, Bonnin HY, Armingaud P, Jaussent A, Picot MC, Le Bars E, Dupeyron A, Arquizan C, Gelis A, Mottet D. Rehabilitation of the upper arm early after stroke: Video games versus conventional rehabilitation. A randomized controlled trial. Ann Phys Rehabil Med. 2020 May;63(3):173-180. doi: 10.1016/j.rehab.2019.10.009. Epub 2019 Dec 9. PMID 31830535